CLINICAL TRIAL: NCT02394574
Title: Household Air Pollution and Pregnancy Outcome
Acronym: HAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 12-1460
Record Dates: First submitted 2015-03-13; First posted 2015-03-20 (Estimated); Last update posted 2024-10-16 (Actual); Status verified 2022-12

CONDITIONS: Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clean Cookstove (Active Comparator): Subjects will use ethanol stoves using bioethanol
  Interventions: Other: Clean Cookstove
- Traditional Cookstove (Other): Subjects will use traditional firewood or kerosine cookstove and receive education on how to reduce air pollution exposures
  Interventions: Other: Traditional Cookstove

INTERVENTIONS:
Other: Clean Cookstove — Ethanol
  Arms: Clean Cookstove
Other: Traditional Cookstove — Firewood / Kerosene
  Arms: Traditional Cookstove

SUMMARY:
Exposure to Household air pollution (HAP) from burning biomass fuels is responsible for an estimated 2.5 million premature deaths and 3.7% of the loss of disability-adjusted life years (DALY) every year in developing countries.52-54 Of all environmental risks, such as unsafe water, poor sanitation, climate change and lead exposure, HAP accounts for the most mortality and DALY.55 Despite the magnitude of the problems associated with HAP, research on its health effects has been hindered by lack of accurate data on exposure and health outcomes. There are few studies available that report HAP exposures and development of adverse pregnancy outcomes from households using biomass fuels.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who present to the hospital
* Who cook exclusively with either kerosene or firewood
* Before the fourteenth week of pregnancy as determined by ultrasound imaging

Exclusion Criteria:

* Smoking women or women with smoking family members
* Women with a high-risk pregnancy defined as:

  * Women with uncontrolled hypertension
  * Women greater than 35 years old carrying their first child
  * Women having triplets or more
  * Women who have had a previous C-section
  * Women carrying babies with fetal abnormalities or as determined by the obstetrician.

Max Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 307 (Actual)
Dates: Start 2012-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Adverse Pregnancy Outcomes | At birth
  (first trimester miscarriages, intrauterine growth retardation, low birth weight (300gm less weight in controls relative to intervention group, premature deliveries (deliveries before 37 weeks of pregnancy) and still births.

SECONDARY OUTCOMES:
Reduction in personal exposure to PM2.5, CO and PAH | At birth
  Reduction in personal exposure to PM2.5, CO and PAH in the Ethanol intervention group relative to the control (kerosene/firewood) group

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Olopade, MD, Principal Investigator — University of Chicago
Locations (1):
- College of Medicine. University of lbadan, Ibadan, Ibadan, Nigeria

REFERENCES:
- [Derived] Deji-Abiodun O, Adedokun B, Alexander D, Dutta A, Ibigbami T, Olamijulo J, Adepoju D, Adekunle S, Ojengbede O, Olopade CO. Impact of prenatal maternal psychological distress on fetal biometric parameters in household air pollution-exposed Nigerian women. PLoS One. 2022 Jul 28;17(7):e0272053. doi: 10.1371/journal.pone.0272053. eCollection 2022. PMID 35901049
- [Derived] Dutta A, Alexander D, Karrison T, Morhasson-Bello O, Wilson N, Atalabi OM, Adu D, Ibigbami T, Adekunle S, Adepoju D, Olamijulo J, Akinwunmi O, Afolabi OS, Deji-Abiodun O, Adedokun B, Aschebrook-Kilfoy B, Ojengbede O, Olopade CO. Household air pollution, ultrasound measurement, fetal biometric parameters and intrauterine growth restriction. Environ Health. 2021 Jun 23;20(1):74. doi: 10.1186/s12940-021-00756-5. PMID 34187482
- [Derived] Alexander D, Northcross A, Wilson N, Dutta A, Pandya R, Ibigbami T, Adu D, Olamijulo J, Morhason-Bello O, Karrison T, Ojengbede O, Olopade CO. Randomized Controlled Ethanol Cookstove Intervention and Blood Pressure in Pregnant Nigerian Women. Am J Respir Crit Care Med. 2017 Jun 15;195(12):1629-1639. doi: 10.1164/rccm.201606-1177OC. PMID 28081369